CLINICAL TRIAL: NCT05741177
Title: Studio Osservazionale, Prospettico, Multicentrico, No-profit Sull' utilità Dell' ECOgrafia Pleuro-polmonare Nella Gestione Delle BRONchioliti Nella Popolazione Pediatrica di età ≤12 Mesi - ECO-BRON
Brief Title: Lung Ultrasound in Bronchiolitis
Acronym: ECOBRON
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID 2021
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- bronchiolitis: children with bronchiolitis
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — lung ultrasound score

SUMMARY:
prospective assessment of lung ultrasound score in children with different severities of bronchiolitis

ELIGIBILITY:
Inclusion Criteria:

* children with bronchiolitis

Exclusion Criteria:

* children with bronchiolitis and comorbidities

Ages: 0 Months to 12 Months | Sex: All
Age Groups: Child
Study Population: Inclusion Criteria:
  * children with bronchiolitis
  Exclusion Criteria:
  * children with bronchiolitis and comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
lung ultrasound score predict bronchiolitis severity | 1 year
  lung ultrasound score predict bronchiolitis severity

CONTACTS AND LOCATIONS:
Locations (1):
- Gemelli Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No